CLINICAL TRIAL: NCT05682131
Title: South China Children Cancer Group - Relapsed-Acute Lymphoblastic Leukemia 2022 Protocol
Acronym: SCCCG-R-ALL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Zhujiang Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Guangzhou First People's Hospital (Other); Huizhou Municipal Central Hospital (Other); First Affiliated Hospital of Shantou University Medical College (Other); Zhongshan People's Hospital, Guangdong, China (Other); Zhongshan Bo Ai Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); LiuZhou People's Hospital (Other); Second Xiangya Hospital of Central South University (Other); Hainan People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYSKY-2022-201-02
Record Dates: First submitted 2023-01-02; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Arsenic Trioxide; Childhood ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Oral placebo was added to conventional chemotherapy
  Interventions: Combination Product: Conventional chemotherapy
- Experimental Group (Experimental): Oral RIF was added to conventional chemotherapy
  Interventions: Drug: Realgar Indigo naturalis formula; Combination Product: Conventional chemotherapy

INTERVENTIONS:
Drug: Realgar Indigo naturalis formula — Realgar Indigo naturalis formula was used in the induction, consolidation and intensive treatment of patients in intermediate or high risk
  Other Names: RIF
  Arms: Experimental Group
Combination Product: Conventional chemotherapy — conventional chemotherapy

SUMMARY:
In recent years, the prognosis of pediatric relapsed ALL patients has improved, but the 5-year OS of patients with first recurrence is still less than 50%. A number of in vitro studies have shown that arsenic trioxide (ATO) can selectively inhibit the growth and induce apoptosis in a variety of leukemia cell lines, suggesting that ATO as a synergist combined with other common chemotherapy drugs may provide a new target for the treatment of relapsed ALL. Realgar Indigo naturalis formula is a compound traditional Chinese medicine preparation developed in China. The main component of realgar is arsenic tetrasulfide (As4S4), which can produce similar pharmacological effects to ATO. Based on the R3 protocol, this study plans to perform a double-blind randomized controlled trial, and to randomly combine compound Huangdai tablets with compound Huangdai tablets in the treatment of intermediate and high risk ALL children, in order to improve the MRD negative rate after induction therapy in this group of children, which may provide a new method for the clinical treatment of relapsed ALL.

DETAILED DESCRIPTION:
In recent years, the prognosis of pediatric relapsed ALL patients has improved, but the 5-year OS of patients with first recurrence is still less than 50%, and the prognosis of children with intermediate and high risk is even worse, so there is an urgent need to explore new and effective treatment methods. A number of in vitro studies have shown that arsenic trioxide (ATO), which is safe and effective in the treatment of APL, can selectively inhibit the growth and induce apoptosis in a variety of leukemia cell lines, suggesting that ATO as a synergist combined with other common chemotherapy drugs may provide a new target for the treatment of relapsed ALL. Realgar Indigo naturalis formula is a compound traditional Chinese medicine preparation developed in China. The main component of realgar is arsenic tetrasulfide (As4S4), which can produce similar pharmacological effects to ATO. The UK ALL R3 protocol is an advanced and mature clinical trial. The results showed that the MRD negative rate after induction chemotherapy and the 2-year DFS of traditional chemotherapy ±HSCT in children with intermediate and high risk did not reach 50%. Based on the R3 protocol, this study plans to perform a double-blind randomized controlled trial, and to randomly combine compound Huangdai tablets with compound Huangdai tablets in the treatment of intermediate and high risk ALL children, in order to improve the MRD negative rate after induction therapy in this group of children, which may provide a new method for the clinical treatment of relapsed ALL.

ELIGIBILITY:
Inclusion Criteria:

* B or T cell type;
* the first recurrence;
* the risk stratification was medium or high risk.

Exclusion Criteria:

* mature B cell leukemia;
* acute mixed phenotype leukemia;
* patients with positive BCR/ABL fusion gene;
* the second tumor
* definite CML blast crisis;
* ALL with Down's syndrome.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2027-09-27 (Estimated); Study Completion 2030-09-27 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | from diagnosis, an average of 7 weeks
  Complete response rate after induction treatment in two groups

CONTACTS AND LOCATIONS:
Overall Officials: Xin Y Chen, Doctoral, Study Chair — Medical Ethics Committee of Sun Yat-sen Memorial Hospital of Sun Yat-sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No